CLINICAL TRIAL: NCT00443105
Title: Topical Tacrolimus 0.03% Ointment for Intractable Allergic Conjunctivitis: An Open Label Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050321
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2007-03-05 (Estimated); Status verified 2006-12

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Tacrolimus; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tacrolimus 0.03% ointment (Protopic)

SUMMARY:
The purpose of this study is to determine the efficacy, tolerance and safety of tacrolimus 0.03% ointment in the treatment of intractable allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included if they were > 5 years old and suffered from intractable allergic conjunctivitis

Exclusion Criteria:

* pregnancy or breastfeeding,history of herpetic eye disease,transplant patients concomitant administration of drugs inhibiting cytochrome CYP3A4, hypersensitivity to macrolides

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: David Zadok, MD, Principal Investigator — Assaf Harofeh Medical Center, Tel Aviv University
Locations (1):
- Assaf Harofeh Medical Center, Department of Ophthalmology, Ẕerifin, Israel